CLINICAL TRIAL: NCT00005194
Title: Insulin and Biogenic Amines in Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1073; R01HL037871 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases; Obesity; Myocardial Infarction; Insulin Resistance
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases; Obesity; Myocardial Infarction; Insulin Resistance

SUMMARY:
To determine the role played by insulin and biogenic amines in obesity-related hypertension and cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

The Normative Aging Study (NAS) is a multidisciplinary longitudinal study of aging established by the Veterans Adminstration in 1963. Six thousand male volunteers from the Greater Boston area were screened for acceptance into the study according to laboratory, clinical, radiologic and electrocardiographic criteria. Volunteers who had a history or presence of such chronic conditions as heart disease, diabetes, cancer, peptic ulcer, gout or recurrent asthma, bronchitis, or sinusitis were not admitted to the study. Also disqualified were those with either systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg. Acceptable conditions included childhood diseases such as rheumatic fever or kidney infection that had not precluded prior military service, as well as hepatitis, malaria, jaundice or anemia, so long as no sequelae were present and functions were intact. Eventually, 2,280 men were accepted into the NAS, ranging in age from 21-81 years with a mean of 42 years. Participants were enrolled and received their first medical examination between 1963 and 1968. Subsequently, men 51 years of age or under have reported for medical examinations every five years. After age 51 they have reported every three years. In 1986, A total of 1,894 subjects remained under active observation with 756 or 33.2 percent being over age 65. The study tested the hypothesis that dietary intake and genetic factors predispose to the development of obesity. Obesity, particularly abdominal obesity characterized by a high waist/hip ratio, is associated with insulin resistance and hyperinsulinemia. The hyperinsulinemia stimulates the sympathetic nervous system and influences the peripheral dopaminergic and serotoninergic systems with the development of hypertension and coincident cardiovascular disease. The study was funded as a result of a Request for Applications for Research in Nutrition and Cardiovascular Disease released in 1986.

DESIGN NARRATIVE:

There were three studies. In the first study, the entire 1,894 subjects of the Normative Aging Study of the Veterans Administration were used. The study was a cross-sectional and longitudinal investigation of the influence of diet and obesity on the production of hyperinsulinism and increased levels of catecholamines, and the relationship of these intermediate outcomes to cardiovascular end points, namely postural change in blood pressure and occurrence of myocardial infarction. Subsets of subjects from the upper and lower quartiles of body mass index and from the upper and lower quartiles of waist/hip ratios were used in the second and third studies.

The second study was cross-sectional and explored the interactions of insulin resistance, sympathetic nervous system activity and cardiovascular function in 80 individuals.

The third study was also cross-sectional, and using the same stratified subsets of subjects, characterized nutrient effects on renal function, particularly sodium excretion and renal amine production.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-09; Study Completion 1991-08 (Actual)

REFERENCES:
- [Background] Landsberg L. Diet, obesity and hypertension: an hypothesis involving insulin, the sympathetic nervous system, and adaptive thermogenesis. Q J Med. 1986 Dec;61(236):1081-90. No abstract available. PMID 3310065
- [Background] Landsberg L. Insulin and hypertension: lessons from obesity. N Engl J Med. 1987 Aug 6;317(6):378-9. doi: 10.1056/NEJM198708063170609. No abstract available. PMID 3299098
- [Background] Krieger DR, Landsberg L. Mechanisms in obesity-related hypertension: role of insulin and catecholamines. Am J Hypertens. 1988 Jan;1(1):84-90. doi: 10.1093/ajh/1.1.84. PMID 3285861
- [Background] Landsberg L, Krieger DR. Obesity, metabolism, and the sympathetic nervous system. Am J Hypertens. 1989 Mar;2(3 Pt 2):125S-132S. doi: 10.1093/ajh/2.3.125s. PMID 2647103
- [Background] Landsberg L. Obesity, metabolism, and hypertension. Yale J Biol Med. 1989 Sep-Oct;62(5):511-9. PMID 2697985
- [Background] Troisi RJ, Weiss ST, Segal MR, Cassano PA, Vokonas PS, Landsberg L. The relationship of body fat distribution to blood pressure in normotensive men: the normative aging study. Int J Obes. 1990 Jun;14(6):515-25. PMID 2401588
- [Background] Landsberg L. Insulin resistance, energy balance and sympathetic nervous system activity. Clin Exp Hypertens A. 1990;12(5):817-30. doi: 10.3109/10641969009073502. PMID 2208753
- [Background] Landsberg L. The sympathoadrenal system, obesity and hypertension: an overview. J Neurosci Methods. 1990 Sep;34(1-3):179-86. doi: 10.1016/0165-0270(90)90056-l. PMID 2259240
- [Background] Sparrow D, O'Connor GT, Young JB, Rosner B, Weiss ST. Relationship of urinary serotonin excretion to cigarette smoking and respiratory symptoms. The Normative Aging Study. Chest. 1992 Apr;101(4):976-80. doi: 10.1378/chest.101.4.976. PMID 1372851
- [Background] Cassano PA, Rosner B, Vokonas PS, Weiss ST. Obesity and body fat distribution in relation to the incidence of non-insulin-dependent diabetes mellitus. A prospective cohort study of men in the normative aging study. Am J Epidemiol. 1992 Dec 15;136(12):1474-86. doi: 10.1093/oxfordjournals.aje.a116468. PMID 1288277
- [Background] Hu H, Sparrow D, Weiss S. Association of serum albumin with blood pressure in the normative aging study. Am J Epidemiol. 1992 Dec 15;136(12):1465-73. doi: 10.1093/oxfordjournals.aje.a116467. PMID 1288276
- [Background] Troisi R, Willett WC, Weiss ST. Trans-fatty acid intake in relation to serum lipid concentrations in adult men. Am J Clin Nutr. 1992 Dec;56(6):1019-24. doi: 10.1093/ajcn/56.6.1019. PMID 1442652
- [Background] Young JB, Troisi RJ, Weiss ST, Parker DR, Sparrow D, Landsberg L. Relationship of catecholamine excretion to body size, obesity, and nutrient intake in middle-aged and elderly men. Am J Clin Nutr. 1992 Nov;56(5):827-34. doi: 10.1093/ajcn/56.5.827. PMID 1415000
- [Background] Landsberg L, Troisi R, Parker D, Young JB, Weiss ST. Obesity, blood pressure, and the sympathetic nervous system. Ann Epidemiol. 1991 May;1(4):295-303. doi: 10.1016/1047-2797(91)90040-j. PMID 1669511
- [Background] Cassano PA, Segal MR, Vokonas PS, Weiss ST. Body fat distribution, blood pressure, and hypertension. A prospective cohort study of men in the normative aging study. Ann Epidemiol. 1990 Oct;1(1):33-48. doi: 10.1016/1047-2797(90)90017-m. PMID 1669488
- [Background] Troisi RJ, Heinold JW, Vokonas PS, Weiss ST. Cigarette smoking, dietary intake, and physical activity: effects on body fat distribution--the Normative Aging Study. Am J Clin Nutr. 1991 May;53(5):1104-11. doi: 10.1093/ajcn/53.5.1104. PMID 1850574
- [Background] Troisi RJ, Weiss ST, Parker DR, Sparrow D, Young JB, Landsberg L. Relation of obesity and diet to sympathetic nervous system activity. Hypertension. 1991 May;17(5):669-77. doi: 10.1161/01.hyp.17.5.669. PMID 2022410
- [Background] Landsberg L. Obesity-related hypertension and the insulin resistance syndrome. Trans Am Clin Climatol Assoc. 1995;106:69-75; discussion 75-6. No abstract available. PMID 7483180
- [Background] Landsberg L. Pathophysiology of obesity-related hypertension: role of insulin and the sympathetic nervous system. J Cardiovasc Pharmacol. 1994;23 Suppl 1:S1-8. PMID 7519690
- [Background] Payton M, Hu H, Sparrow D, Weiss ST. Low-level lead exposure and renal function in the Normative Aging Study. Am J Epidemiol. 1994 Nov 1;140(9):821-9. doi: 10.1093/oxfordjournals.aje.a117330. PMID 7977292
- [Background] Ward KD, Sparrow D, Vokonas PS, Willett WC, Landsberg L, Weiss ST. The relationships of abdominal obesity, hyperinsulinemia and saturated fat intake to serum lipid levels: the Normative Aging Study. Int J Obes Relat Metab Disord. 1994 Mar;18(3):137-44. PMID 8186810
- [Background] Ward KD, Sparrow D, Landsberg L, Young JB, Vokonas PS, Weiss ST. The relationship of epinephrine excretion to serum lipid levels: the Normative Aging Study. Metabolism. 1994 Apr;43(4):509-13. doi: 10.1016/0026-0495(94)90085-x. PMID 8159112
- [Background] Payton M, Hu H, Sparrow D, Young JB, Landsberg L, Weiss ST. Relation between blood lead and urinary biogenic amines in community-exposed men. Am J Epidemiol. 1993 Nov 15;138(10):815-25. doi: 10.1093/oxfordjournals.aje.a116785. PMID 8237970
- [Background] Landsberg L, Young JB. Sympathoadrenal activity and obesity: physiological rationale for the use of adrenergic thermogenic drugs. Int J Obes Relat Metab Disord. 1993 Feb;17 Suppl 1:S29-34. PMID 8384176
- [Background] Parker DR, Weiss ST, Troisi R, Cassano PA, Vokonas PS, Landsberg L. Relationship of dietary saturated fatty acids and body habitus to serum insulin concentrations: the Normative Aging Study. Am J Clin Nutr. 1993 Aug;58(2):129-36. doi: 10.1093/ajcn/58.2.129. PMID 8338037
- [Background] Young JB, Macdonald IA. Sympathoadrenal activity in human obesity: heterogeneity of findings since 1980. Int J Obes Relat Metab Disord. 1992 Dec;16(12):959-67. PMID 1335975
- [Background] Landsberg L. Obesity and hypertension: experimental data. J Hypertens Suppl. 1992 Dec;10(7):S195-201. PMID 1291654
- [Background] Landsberg L. Hyperinsulinemia: possible role in obesity-induced hypertension. Hypertension. 1992 Jan;19(1 Suppl):I61-6. doi: 10.1161/01.hyp.19.1_suppl.i61. PMID 1730456
- [Background] Daly PA, Landsberg L. Pathogenesis of hypertension in NIDDM: lessons from obesity. J Hum Hypertens. 1991 Aug;5(4):277-85. No abstract available. PMID 1956026
- [Background] Daly PA, Landsberg L. Hypertension in obesity and NIDDM. Role of insulin and sympathetic nervous system. Diabetes Care. 1991 Mar;14(3):240-8. doi: 10.2337/diacare.14.3.240. PMID 2044439
- [Background] Manning WJ, Shannon RP, Santinga JA, Parker JA, Gervino EV, Come PC, Wei JY. Reversal of changes in left ventricular diastolic filling associated with normal aging using diltiazem. Am J Cardiol. 1991 Apr 15;67(9):894-6. doi: 10.1016/0002-9149(91)90628-x. No abstract available. PMID 2011992
- [Background] Lipsitz LA, Jonsson PV, Marks BL, Parker JA, Royal HD, Wei JY. Reduced supine cardiac volumes and diastolic filling rates in elderly patients with chronic medical conditions. Implications for postural blood pressure homeostasis. J Am Geriatr Soc. 1990 Feb;38(2):103-7. doi: 10.1111/j.1532-5415.1990.tb03469.x. PMID 2299113